CLINICAL TRIAL: NCT07358026
Title: EARLY-PREG: A Preconception, Longitudinal, Bidirectional, and Counterfactual Cohort Study of Women Seeking Pregnancy, Designed to Investigate Maternal-Embryonic Molecular Interactions During the Pre- and Peri-implantation Windows
Brief Title: EARLY-PREG: A Preconception Cohort Study Based on Counterfactuals to Study Maternal-Embryonic Molecular Interactions
Acronym: EARLY-PREG
Status: Recruiting | Type: Observational
Sponsor: MELISA Institute Genomics & Proteomics Research SpA (Industry)
Responsible Party: Principal Investigator, Elard Koch, PhD, Head of research, MELISA Institute Genomics & Proteomics Research SpA
Other Study IDs: 17-03-06; MEL109112011, MEL109112011R4 (Other Grant/Funding Number: Fundacion de investigacion san Ramon (FISAR)); MEL109112011R5, MEL131032017R1 (Other Grant/Funding Number: Fundacion de investigacion san Ramon (FISAR)); MEL205062018, REH042024-01 (Other Grant/Funding Number: Fundacion de investigacion san Ramon (FISAR))
Record Dates: First submitted 2026-01-08; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Early Pregnancy; Early Pregnancy Loss; Childbirth; Healthy; Pregnancy
Keywords: longitudinal study; counterfactual design; embryo-mother crosstalk; biorepository; maternal fluids; menstrual cycle; preconception open cohort
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Saliva, urine, blood, cervicovaginal fluid, cervical brushings, umbilical cord blood and placenta.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CONCEPTION CYCLE: Conception cycle refers to the menstrual cycle in which the ovum is fertilised, leading to pregnancy. Confirmation of a conception cycle requires beta-hCG levels above the clinical threshold for a positive pregnancy test, which is determined in peripheral venous blood on the 14th day post-ovulation.
  Interventions: Other: EMBRYO EXPOSURE
- NON-CONCEPTION CYCLE: Non-conception cycle refers to a menstrual cycle in which pregnancy does not occur. When referring to the same individual, it is, by definition, considered the counterfactual to the conception cycle described above. Confirmation of a non-conception cycle requires a clinically negative beta-hCG test, determined in peripheral venous blood on the 14th day post-ovulation. This cycle is characterised by the absence of a clinical pregnancy.

INTERVENTIONS:
Other: EMBRYO EXPOSURE — The counterfactual design of EARLY-PREG enables the comparison of the systemic and localised physiological effects associated with embryo appearance and implantation in an individual (the factual) against the physiological state of the same individual without experiencing pregnancy (the counterfactual).
  Groups: CONCEPTION CYCLE

SUMMARY:
EARLY-PREG is an open-cohort clinical study with a preconception, longitudinal, bidirectional and counterfactual design. The aim of this cohort is to investigate the proteomic signatures of maternal-embryonic communication by interrogating a growing biorepository of maternal fluids and tissues collected during the first two weeks after fertilisation.

Participants in the EARLY-PREG cohort consist of healthy couples seeking pregnancy, as well as women who are not seeking to conceive. The three main outcomes in the cohort are defined according to menstrual cycles in which conception is achieved and those in which conception is not achieved. Their clinical definitions are as follows:

* Pregnancy with a full-term live birth refers to the cycle in which the ovum is fertilised, leading to pregnancy, with beta-hCG levels above the clinical threshold for a positive pregnancy test.
* Early pregnancy loss refers to a miscarriage up to 12 6/7 weeks.
* Non-pregnancy refers to a menstrual cycle in which conception does not occur, confirmed by a clinically negative beta-hCG test. When referring to the same individual, this is, by definition, considered the counterfactual to the corresponding conception cycle.

DETAILED DESCRIPTION:
Successful pregnancy depends on a coordinated exchange of signals between the early embryo and the mother. This complex process begins immediately after fertilisation, during the pre-implantation period. Although it plays a critical role in preparing the maternal environment for pregnancy, the mechanisms behind this communication remain incompletely understood.

The unique 'dialogue' between the embryo and the mother is a bidirectional exchange known as embryo-maternal crosstalk. Evidence indicates that this interaction, mediated by molecular signals present in uterine fluid, supports appropriate embryo implantation and modulates the maternal immune system to facilitate tolerance of the developing embryo.

To date, the majority of knowledge in this field has been derived from animal models and in vitro studies, which may not fully represent the physiology of spontaneous human conception. The EARLY-PREG preconception open cohort has been established to address this gap by characterising embryo-maternal crosstalk in vivo. This study follows healthy women who are trying to become pregnant, following them from before conception through the first two weeks of a natural conception, with continued follow-up into pregnancy and childbirth.

Daily collection of a range of biological samples - including saliva, urine, blood, cervicovaginal fluid and cervicovaginal brushings - is undertaken during key phases of the menstrual cycle. These samples are processed, preserved and stored in a dedicated biorepository for subsequent analysis using omics-based approaches.

ELIGIBILITY:
Inclusion criteria:

* being between 18 and 40 years of age
* not being pregnant
* normal colposcopy
* body mass index (BMI) between 18 and 29
* regular menstrual cycles (21-35 days)
* absence of chronic diseases (hypertension, diabetes mellitus, cancer, depression, personality disorder, thyroid pathology, polycystic ovary syndrome, or hyperprolactinemia).
* If seeking pregnancy, they were included if their partners were males between 18 and 40 years old, without pathologies (diabetes mellitus, depression, personality disorder, or cancer), were not taking chronic medication, without erectile disorders, BMI between 18 and 29.9, moderate alcohol use, and with no recreational drug use.

Exclusion criteria:

* pregnant women
* history of alcoholism
* infertility treatment
* endometriosis
* pelvic inflammatory disease
* pelvic surgery
* allergy to latex or silicone
* If seeking pregnancy, they were excluded if their partners were working in contact with pesticides, or with history of erectile dysfunction, or history of mumps in adulthood, or with chronic diseases, or with psychological problems.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women visiting gynaecologists, and midwives in private practices, public hospitals, and Family Health Centres (CESFAMs) in the Biobio region of Chile.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of menstrual cycles leading to full-term pregnancies | From enrollment for up to six menstrual cycles (each cycle ranges from 21-35 days) or until pregnancy resulting in live birth, whichever occurs first.
  This outcome refers to the menstrual cycle in which the ovum is fertilised, leading to pregnancy with a full term live birth. The conception cycle requires beta-hCG levels above the clinical threshold for a positive pregnancy test, which is determined in peripheral venous blood on the 14th day post-ovulation.
Number of menstrual cycles not leading to pregnancy | From enrollment for up to six menstrual cycles (each cycle ranges from 21-35 days) or until pregnancy occurs, whichever occurs first.
  This outcome refers to a menstrual cycle in which pregnancy does not occur. When referring to the same individual, it is, by definition, considered the counterfactual to the conception cycle described above. A non-conception cycle is confirmed by a clinically negative beta-hCG test, which is determined in peripheral venous blood on the 14th day post-ovulation. This cycle is characterised by the absence of a clinical pregnancy.
Number of menstrual cycles leading to early pregnancy loss | From the time beta-hCG levels rise above the clinical threshold for a positive pregnancy test until a miscarriage occurring up to 12 6/7 weeks.
  This outcome refers to the menstrual cycle in which the ovum is fertilised, leading to a miscarriage until 12 6/7 weeks. The conception cycle requires beta-hCG levels above the clinical threshold for a positive pregnancy test, which is determined in peripheral venous blood on the 14th day post-ovulation.

CONTACTS AND LOCATIONS:
Overall Officials: Elard S Koch, Study Director — MELISA Institute Genomics & Proteomics Research SpA
Locations (1):
- Clínica Sanatorio Alemán, Chiguayante, Chile

IPD SHARING:
Plan to Share IPD: Yes
All IPD information underlying the results of a publication will be shared with the sole exception of sensitive information that could reveal a person's identity.
Supporting Information: Study Protocol
Time Frame: January 2027 - December 2028
Access Criteria: The protocol data and results will be deposited in appropriate public repositories.

REFERENCES:
- See also: MELISA Institute — http://www.melisainstitute.org